CLINICAL TRIAL: NCT06358274
Title: Nutritional and Metabolic Dynamics of Thru-Hiking: A Longitudinal Study on the Colorado Trail
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: MED-2024-32848
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Thru-hiking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood collected for a blood lipid panel
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- thru-hiking on the Colorado Trail: Thru-hikers planning to embark on the Colorado Trail are recruited through the Colorado Trail Foundation community page and email newsletter, ensuring a sample population representative of those undertaking this challenging endeavor.
  Participants will be tracked over time to assess changes in their metabolic health and dietary habits.
  Interventions: Other: Thru-hiking

INTERVENTIONS:
Other: Thru-hiking — planning to embark on the Colorado Trail

SUMMARY:
Thru-hiking the Colorado Trail presents distinct challenges owing to its diverse landscapes and high altitudes. The study aims to delve into the physiological and nutritional facets of extended wilderness trekking among thru-hikers. Activities encompass participant recruitment from the Colorado Trail Foundation community, baseline and post-trail assessments including blood lipid panel analysis and anthropometric measurements, data collection during the trail period involving recording daily mileage, exertion levels, and dietary intake, rigorous statistical analysis to explore correlations among various parameters, and adherence to ethical considerations including obtaining formal approval and ensuring informed consent procedures are followed to safeguard participants' rights and privacy. Through this endeavor, the study seeks to offer insights into the metabolic responses and cardiovascular implications associated with thru-hiking, shedding light on the interplay between diet, lifestyle factors, and metabolic health in challenging environments.

The specific aims include examining the metabolic responses and cardiovascular implications associated with thru-hiking, exploring correlations between dietary intake and blood lipid profiles, and elucidating the interplay between lifestyle factors and metabolic health in demanding environments. This study is not limited to program evaluation, quality assurance, or improvement activities within a specific department or setting but rather seeks to contribute to scientific knowledge and inform evidence-based recommendations for individuals engaging in thru-hiking or similar high-intensity activities.

ELIGIBILITY:
Inclusion Criteria:

* Thru-Hikers on the Colorado Trail:
* Individuals planning to commence their thru-hiking journey on the Colorado Trail in early July.

Residence:

* Participants must reside in northern Colorado.
* Thru-Hiking History
* Participants must not have completed another thru-hike in the past 6 months.
* Informed Consent
* Individuals interested in participating in the study must provide informed consent.

Exclusion Criteria:

* Individuals who have completed another thru-hike in the past 6 months
* children below the age of majority, pregnant women, fetuses, and neonates
* prisoners, adults lacking the capacity to consent or with fluctuating capacity, non-English speakers, and illiterate individuals
* employees or students of the researcher
* individuals from undervalued or disenfranchised social groups
* Active members of the military, including Department of Defense (DoD) personnel
* individuals in stressful situations, those disadvantaged in social goods and services and individuals with serious health conditions lacking standard treatments
* those with a fear of negative consequences for not participating and individuals facing circumstances increasing vulnerability to coercion or exploitation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals hiking The Colorado Trail in its entirety in summer 2024. Excluded are those having hiked another thru-hike 6 months prior.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
blood lipid panel: total cholesterol | baseline and 2 days post-hike
  changes in total cholesterol levels from baseline to within 2 days of completing the Colorado Trail.
blood lipid panel: high-density lipoprotein (HDL) | baseline and 2 days post-hike
  changes in HDL levels from baseline to within 2 days of completing the Colorado Trail.
blood lipid panel: low-density lipoprotein (LDL) | baseline and 2 days post-hike
  changes in LDL levels from baseline to within 2 days of completing the Colorado Trail.
blood lipid panel: triglycerides | baseline and 2 days post-hike
  changes in triglycerides levels from baseline to within 2 days of completing the Colorado Trail.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Selinsky, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States